CLINICAL TRIAL: NCT00137696
Title: Immunogenicity of Inactivated Polio Vaccine in Puerto Rico; A Comparative Cohort Study of Two Vaccination Schedules
Brief Title: Comparison of Immune Response Using 2 Vaccination Schedules Using Inactivated Polio Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: San Lucas Hospital, Ponce, Puerto Rico (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: CDC-NIP-3436; 020918-YY (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Poliomyelitis
Keywords: polio; vaccine; immunogenicity
MeSH Terms: conditions — Poliomyelitis | interventions — Vaccination; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cohort A-WHO/EPI Schedule (Experimental): Received IPV at ages 6, 10, and 14 weeks (this schedule is also approved for use in the United States if an accelerated schedule is needed.
  Interventions: Biological: Vaccination with inactivated polio vaccine; Procedure: Collection of serum
- Cohort A-US Schedule (Active Comparator): Received IPV at ages 8, 16, and 24 weeks.
  Interventions: Biological: Vaccination with inactivated polio vaccine; Procedure: Collection of serum

INTERVENTIONS:
Biological: Vaccination with inactivated polio vaccine
Procedure: Collection of serum

SUMMARY:
As poliovirus eradication progresses rapidly, strategies to discontinue oral poliovirus vaccination need to be established. One strategy would be to use inactivated poliovirus vaccine (IPV) transitionally, and this has already occurred in the United States. It is not clear, however, if 3 doses of IPV provide sufficient immunogenicity when administered according to World Health Organization (WHO)/Expanded Programme on Immunization (EPI) schedule in a tropical, developing area where no wild-poliovirus circulates.

Puerto Rico will be the study site for this randomized clinical trial. Healthy infants will be identified at birth in a hospital-system, enrolled within 4 weeks of birth, and randomized into one of two arms: United States of America (U.S.A.) schedule (8, 16, 24 weeks/2, 4, 6 months) or WHO schedule (6, 10, 14 weeks). Both groups will receive IPV at visits 1, 2 and 3. Infants will receive all age-appropriate EPI childhood vaccinations along with IPV, to decrease confusion and inconvenience to the parent. Serum will be collected twice, at visit 1 and visit 4 (30-45 days after IPV-3), to measure antibody titers. Sera will be measured for neutralizing antibodies at the Centers for Disease Control (CDC). Based on the lowest seroconversion rate estimate of 85%, and to have a probability of .80 that the estimate from this study is in error by no more than 10%, the investigators will need to enroll 220 infants in each arm. To compensate for attrition and retain statistical power, the investigators plan to enroll up to 250 infants in each arm. This study is expected to require at least 20 months to complete. Results will provide valuable and timely information applicable to global polio eradication efforts. Any participant found not to be protected after 3 doses of IPV will be given a booster at 9-12 months. Results will provide valuable and timely information applicable to global polio eradication efforts.

DETAILED DESCRIPTION:
The proposed study will be a prospective, randomized clinical trial of the immunogenicity of IPV among two groups of infants using different immunization schedules (WHO/EPI and US).

Study will begin with an enrollment period up to 10 months. All infants born at San Lucas Hospital will be eligible unless otherwise excluded. The study will continue until 10 months after the last infant is enrolled. There will be four or five study visits, depending on the cohort.

Study Population:

Infants will be identified at birth at San Lucas Hospital; all babies born during the enrollment period at the selected hospital will be considered eligible. Mothers will be approached in the hospital by the study -nurse after infant's birth and be informed about the study. Inclusion and exclusion criteria will be assessed at this time and if the mother agrees to the study, informed consent will be obtained.

Randomization will be based on what day the baby was born. Even days will be assigned to the WHO schedule and odd days to the US schedule. The mother will be told which cohort the infant is in and given an immunization card with dates that the infant is to return to receive vaccinations. The card will also include study contact phone numbers.

The study will be implemented through the Ponce School of Medicine at San Lucas Hospital in Ponce Puerto Rico. This teaching hospital has a 24 bed well-baby nursery where approximately 150 babies are born per month.

Interventions:

To avoid confusion, inconvenience and error, and to limit differences among participants, diphteria-tetanus-acellular pertussis (DTaP), Haemophilus influenzae type B (Hib), pneumococcal conjugate vaccine (PCV), and hepatitis B (HepB) (if appropriate) will be administered along with inactivated poliovirus vaccine (IPV) on first 3 visits in both cohorts. Both schedules meet the parameters of Advisory Committee of Immunization Practices (ACIP) (minimum interval at least 4 weeks between doses and minimum age of 6 weeks of age) 2.

Cohort A-WHO/EPI Schedule

Initial Study Visit: Visit 1 will be scheduled for 6 weeks (> 42 days and < 46 days) after birth. Blood will be drawn (sera 1) immediately prior to administration with first dose of IPV and other recommended vaccines. Mother will be reminded of infant's next appointment in 4 weeks.

Study Visit 2: Visit 2 will be scheduled for 4 weeks after last vaccination (> 28 days and < 32 days). The 2nd dose of IPV and other recommended vaccines will be administered at this time. Mother will be reminded of infant's next appointment in 4 weeks.

Study Visit 3: Visit 3 will be scheduled for 4 weeks after last vaccination (> 28 days and < 32 days). The 3rd dose of IPV and other recommended vaccines will be administered at this time. Mother will be reminded of infant's next appointment in 4 weeks.

Study Visit 4: Visit 4 will be scheduled for 4 weeks after last vaccination. A blood sample will be drawn from participant. Study visit should take place no earlier than 28 days since previous vaccination nor later than the 45th day

Study Visit 5: According to ACIP recommendations the 3rd dose of Hepatitis B has to be administered after 6 months of age. For this reason, Visit 5 will be scheduled when the child is 24 weeks of age in order to receive the 3rd dose of Hepatitis B vaccine.

Cohort B-US Schedule

Initial Study Visit: Visit 1 will be scheduled for 8 weeks after birth (> 52 days and < 60 days). Blood will be drawn (sera 1) immediately prior to administration of the first dose of IPV and other recommended vaccines. Mother will be reminded of infant's next appointment in 8 weeks.

Study Visit 2: Visit 2 will be scheduled for 8 weeks after last vaccination (> 52 days and < 60 days). The 2nd dose of IPV and other recommended vaccines will be administered. Mother will be reminded of infant's next appointment in 8 weeks.

Study Visit 3: Visit 3 will be scheduled for 8 weeks after last vaccination (> 52 days and < 60 days). The 3rd dose of IPV and other recommended vaccines will be administered at this time. Mother will be reminded of infant's next appointment in 4 weeks.

Study Visit 4: Visit 4 will be scheduled for 4 weeks after last vaccination. A blood sample will be drawn from participant. Study visit should take place no earlier than 28 days since previous vaccination nor later than the 45th day.

Specimens Collection/Handling:

Blood will be drawn to obtain serum neutralizing antibody titers prior to the first dose of IPV and subsequent to the 3rd dose of IPV. If >= 2% of children in either arm do not respond to any of the 3 types of poliovirus, two additional blood specimens will be offered to test immunity before and after the 4th dose of IPV among non responders.

A minimum of 500 µl will be collected at each bleed preferably via vein using a 23-25 gauge butterfly into a vacutainer tube (heel stick is acceptable if infant is noted to have poor venous access). Specimens will be labeled with a unique identifier and be kept cold (2-8° C), not frozen, until specimen is spun down and sera separated which should be done at end of each day (specimens should not sit out for > 12 hours).

Sera will be aliquoted and batch-stored at -20° C. A batched frozen shipment on dry ice will be made to CDC after Phase 1 (all participant study visits are complete).

Lab Evaluation and Methods:

Sera will be tested for levels of neutralizing antibody titers against poliovirus types 1, 2 and 3 at CDC by means of a modified microneutralization assay 13. Approximately 80 to 100 median tissue culture infective dose (TCID50) of each vaccine virus serotype and serial dilutions of serum (starting at 1:8 and ending at 1:1024) are incubated at 37° C for 2.5 hours before 7.5x103 Hep-2(C) cells are added to the wells. After incubation for 5 days at 37° C, each plate is stained with 0.05% crystal violet in 25% ethyl alcohol, with the optical density in each well measured by a spectrophotometer. Each specimen will be run in triplicate, with the final titer estimated by the method of Spearman-Karber. Seropositivity will be defined as a neutralization titer of greater than 1:8. It is estimated that serology results will be available 60 days after receipt of specimens at CDC.

Analysis:

This study is designed to examine and compare seroconversion in response to IPV given according to the WHO/EPI and US schedules. Our primary interest is to determine whether the seroconversion rate among children receiving the WHO/EPI schedule is no lower than 10% less than the rate among those using the US schedule. To determine the required number of study participants, we will assume that the seroconversion rate using the US schedule will be 85% and we want power of .80 to find a significant difference between the rates if the rate among the WHO/EPI schedule group is 75% or lower. Using a one-tailed test (and realizing that one-sided significance levels are uncommon in epidemiologic studies and give us a confidence level of only 90% and not the standard 95%) based on the normal approximation of the binomial distribution, a sample size of ~220 subjects per arm will satisfy these criteria. To compensate for expected attrition of ~14 % , a goal of 250 infants will be set for each arm.

Study Drug:

IPV is an FDA licensed drug. No investigational drugs are being used for the purpose of this study. No routine vaccinations are being withheld for the purpose of this study. Those participants randomized to the WHO/EPI schedule will receive their vaccines on a different time schedule than they would usually follow in Puerto Rico. However, both schedules meet the parameters of the Advisory Committee of Immunization Practices (ACIP) 2. Because participants will be followed closely for up to 6 months of life, it is likely that they will receive their vaccinations in a more timely manner than they might if not a part of the study. Parents will be given a unique immunization card showing the schedule their infant will follow; all vaccines administered will be recorded. The card will indicate that they are enrolled in a study and list study staff names and contact telephone numbers.

Informed Consent Procedures:

Prior to infant vaccination, parents will be given standard vaccine information statements (VIS) and informed consents in Spanish or English, as they would if they were to immunize their child with their pediatrician or health clinic. Information and risks of all administered vaccines will not be discussed in the study informed consent, as the form would be overwhelmingly long.

Confidentiality:

Confidentiality will be assured by keeping all identifying material in a locked cabinet in a locked office. All personal identifiers will be removed before data and specimens are shipped to CDC. Records will be held confidential to the fullest extent allowed by state and federal laws.

Information collected for this study will include only a minimum degree of sensitive personal information in the form of demographic data. Its disclosure should pose negligible risk to participant and or/parent. Parents will be provided with the usual written information discussing pros and cons on each vaccine to be administered.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 48 hours of age born at San Lucas Hospital during study enrollment period
* Infants with gestational age of > 37 weeks as assessed by neonatologist
* Mother/guardian gives informed consent
* Infant is expected to reside in Puerto Rico for the following 8 months

Exclusion Criteria:

* Mother/guardian does not speak English or Spanish
* Mother/guardian has religious/philosophical objection to immunizations
* Infant has serious chronic or acute health problems that require hospitalization immediately (within 1 day) after birth (assessed by infant not being placed in San Lucas Hospital well-baby clinic)
* Mother expects to travel with infant during study period to a country known to have circulating poliovirus or that uses oral poliovirus vaccine (OPV)

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 473 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Serum collection and antibody titers | 30-45 days after vaccination
  Serum will be collected twice, at visit 1 and visit 4 (30-45 days after IPV-3), to measure antibody titers.

SECONDARY OUTCOMES:
Adverse Events | 7 days after vaccination
  Reports on adverse events will be obtained after each vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo H Dayan, MD, Principal Investigator — Centers for Disease Control and Prevention; Margaret Thorley, MPH, Study Chair — Centers for Disease Control and Prevention; Steve McLaughlin, DV, Study Chair — Centers for Disease Control and Prevention; Mark Pallansch, Study Chair — Centers for Disease Control and Prevention; Yasuhiro Yamamura, PhD, Study Director — Ponce School of Medicine; Nayra Rodriguez, Study Chair — Ponce School of Medicine
Locations (1):
- Ponce School of Medicine, Ponce, Puerto Rico

REFERENCES:
- [Result] Dayan GH, Thorley M, Yamamura Y, Rodriguez N, McLaughlin S, Torres LM, Seda A, Carbia M, Alexander LN, Caceres V, Pallansch MA. Serologic response to inactivated poliovirus vaccine: a randomized clinical trial comparing 2 vaccination schedules in Puerto Rico. J Infect Dis. 2007 Jan 1;195(1):12-20. doi: 10.1086/508427. Epub 2006 Nov 28. PMID 17152004